CLINICAL TRIAL: NCT05542238
Title: The Effect of Acute Exercise on Cardiac Autonomic, Cerebrovascular, and Cognitive Function in Spinal Cord Injury: a Pilot Study
Brief Title: The Effect of Acute Exercise on Cardiac Autonomic, Cerebrovascular, and Cognitive Function in Spinal Cord Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We have enrolled all the required participants for this pilot study.
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Wenjie Ji, PhD student, State University of New York at Buffalo
Allocation: Not Applicable | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00006517-Pilot
Record Dates: First submitted 2022-09-07; First posted 2022-09-15 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injuries; Cardiovascular Abnormalities; Cerebrovascular Disease; Sequelae; Cognitive Impairment
MeSH Terms: conditions — Spinal Cord Injuries; Cardiovascular Abnormalities; Cerebrovascular Disorders; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CON (Active Comparator): Age-and sex-matched healthy controls with exercise intervention
  Interventions: Behavioral: One bout of moderate-intensity sub-maximal aerobic exercise
- SCI (Experimental): Individuals with spinal cord injury
  Interventions: Behavioral: One bout of moderate-intensity sub-maximal aerobic exercise

INTERVENTIONS:
Behavioral: One bout of moderate-intensity sub-maximal aerobic exercise — The intervention is a 20-min acute exercise using arm ergometer

SUMMARY:
The aims of this proposal are to: 1) investigate whether individuals with spinal cord injury (SCI) demonstrate cardiac autonomic, cerebrovascular, and cognitive dysfunctions compared to non-injured age- and sex-matched controls in the following conditions: supine rest and head-up tilt/face-cooling test; 2) examine if autonomic completeness/ incompleteness, physical activity, and psychological distress are predictors for dysfunctions during supine rest and head-up tilt/face cooling conditions in SCI individuals; 3) examine if one bout of moderate-intensity aerobic exercise temporarily improves cardiac autonomic and cerebrovascular functions and thereby improves cognition when in supine rest and head- up tilt/face cooling conditions. The study will include an initial visit and an experimental visit to our lab. Three groups of participants will be included in this study: Group 1, SCI with acute exercise; group 2, SCI with rest-control; and group 3, age- and sex-matched non-injured individuals. Cardiovascular variables, such as heart rate variability, blood pressure variability, and cerebrovascular variables, such as cerebral blood flow velocity and oxygenated hemoglobin, and cognitive performance will be examined. The investigator hypothesizes that individuals with SCI will have impaired cardiac autonomic, cerebrovascular, and cognitive functions compared to the non-injured controls, and an acute exercise can improve those functions. Autonomic completeness/incompleteness, physical activity, and psychological distress are significant factors that predict cardiac autonomic, cerebrovascular, and cognitive functions in individuals with SCI.

ELIGIBILITY:
Inclusion Criteria:

Spinal cord injury group:

* Males or females with chronic SCI (i.e. at least 6 months after the initial injury)
* International Standard for Neurological Classification of SCI (ISNCSCI) A-D
* Neurological level of injury C6 or below
* 18-55 years old
* Proficient in English
* Able to detect middle cerebral artery blood velocity (MCAv) and/or posterior cerebral artery blood velocity (PCAv) signals through TCD

Non-injured controls:

* Males or females without SCI
* 18-55 years old
* Proficient in English
* Able to detect MCAv and/or PCAv signals through TCD

Exclusion Criteria:

* Cardiovascular, pulmonary or respiratory diseases, or diabetes mellitus, any other diseases/disorders affecting cardiac autonomic nervous system, such as glaucoma and attention deficit hyperactivity disorder (ADHD)
* Color Blindness
* Pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Cardiac sympathetic function | During baseline pre the 20-min acute exercise
  Low frequency component of blood pressure variability in mmHg^2
Cardiac parasympathetic function | During baseline pre the 20-min acute exercise
  High frequency component of heart rate variability in mm^2
Cardiac sympathetic function | During face-cooling test pre the 20-min acute exercise
  Low frequency component of blood pressure variability in mmHg^2
Cardiac parasympathetic function | During face-cooling test pre the 20-min acute exercise
  High frequency component of heart rate variability in mm^2
Cardiac sympathetic function | During head-up tilt test pre the 20-min acute exercise
  Low frequency component of blood pressure variability in mmHg^2
Cardiac parasympathetic function | During head-up tilt test pre the 20-min acute exercise
  High frequency component of heart rate variability in mm^2
Cardiac sympathetic function | During cognitive tests pre the 20-min acute exercise
  Low frequency component of blood pressure variability in mmHg^2
Cardiac parasympathetic function | During cognitive tests pre the 20-min acute exercise
  High frequency component of heart rate variability in mm^2
Cardiac sympathetic function | During baseline post the 20-min acute exercise
  Low frequency component of blood pressure variability in mmHg^2
Cardiac sympathetic function | During face-cooling post the 20-min acute exercise
  Low frequency component of blood pressure variability in mmHg^2
Cardiac parasympathetic function | During face-cooling post the 20-min acute exercise
  High frequency component of heart rate variability in mm^2
Cardiac sympathetic function | During head-up tilt test post the 20-min acute exercise
  Low frequency component of blood pressure variability in mmHg^2
Cardiac parasympathetic function | During head-up tilt test post the 20-min acute exercise
  High frequency component of heart rate variability in mm^2
Cardiac sympathetic function | During cognitive tests post the 20-min acute exercise
  Low frequency component of blood pressure variability in mmHg^2
Cardiac parasympathetic function | During cognitive tests post the 20-min acute exercise
  High frequency component of heart rate variability in mm^2
Cerebrovascular functions | During baseline pre the 20-min acute exercise
  Assessed by the middle and posterior cerebral artery velocity in centimeters per second
Cerebrovascular functions | During the face-cooling test pre the 20-min acute exercise
  Assessed by the middle and posterior cerebral artery velocity in centimeters per second
Cerebrovascular functions | During the head-up tilt test pre the 20-min acute exercise
  Assessed by the middle and posterior cerebral artery velocity in centimeters per second
Cerebrovascular functions | During the cognitive tests pre the 20-min acute exercise
  Assessed by the middle and posterior cerebral artery velocity in centimeters per second
Cerebrovascular functions | During baseline post the 20-min acute exercise
  Assessed by the middle and posterior cerebral artery velocity in centimeters per second
Cerebrovascular functions | During the face-cooling test post the 20-min acute exercise
  Assessed by the middle and posterior cerebral artery velocity in centimeters per second
Cerebrovascular functions | During the head-up tilt test post the 20-min acute exercise
  Assessed by the middle and posterior cerebral artery velocity in centimeters per second
Cerebrovascular functions | During the cognitive tests post the 20-min acute exercise
  Assessed by the middle and posterior cerebral artery velocity in centimeters per second
Cerebral oxygenation level | Change from baseline to the cognitive tests pre the 20-min acute exercise
  Cerebral oxygenated hemoglobin in unknown unit
Cerebral oxygenation level | Change from baseline to the cognitive tests post the 20-min acute exercise
  Cerebral oxygenated hemoglobin in unknown unit
Cognitive function | During baseline pre the 20-min acute exercise
  Reaction time in second
Cognitive function | During baseline pre the 20-min acute exercise
  Error made during the cognitive test in number
Cognitive function | During head-up tilt pre the 20-min acute exercise
  Reaction time in second
Cognitive function | During head-up tilt pre the 20-min acute exercise
  Error made during the cognitive test in number
Cognitive function | During baseline post the 20-min acute exercise
  Reaction time in second
Cognitive function | During baseline post the 20-min acute exercise
  Error made during cognitive test in number
Cognitive function | During head-up tilt post the 20-min acute exercise
  Reaction time in second
Cognitive function | During head-up tilt post the 20-min acute exercise
  Error made during the cognitive test in number

CONTACTS AND LOCATIONS:
Overall Officials: Wenjie Ji, MS, Principal Investigator — University at Buffalo
Locations (1):
- Department of Rehabilitation Sciences at University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No